CLINICAL TRIAL: NCT00500383
Title: Breast Cancer Risk Assessment Using Optical Breast Spectroscopy (OBS)
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Mount Sinai Hospital, Canada (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: UHNREB#07-0689-CE; HC#124313
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer Risk; BRCA1; BRCA2; Breast Cancer Susceptibility gene; Optical Transillumination Spectroscopy; Transillumination Breast Spectroscopy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to evaluate if a light based technique, called Optical Breast Spectroscopy (OBS) formerly known as Transillumination Breast Spectroscopy (TiBS), can be used to detect differences in breast tissue between high- and low-risk populations and within the high-risk population between BrCa1 or 2 carriers and non-carriers. These differences may include differences in breast tissue composition and metabolism at time of enrollment into the study (possibly reflecting changes occurring in adolescence) and in the rate of breast tissue change over time (possibly reflecting rate of tissue transformation from normal to ultimately malignant state).

DETAILED DESCRIPTION:
Preliminary data show Optical Breast Spectroscopy (OBS)has the ability to detect tissue differences with various pathologies and age-related changes in breast tissue over a two year period. In the present study, we want to determine whether OBS has the ability to detect optical differences between women who harbor a mutation in the breast cancer susceptibility gene, BrCa1 or BrCa2, and their age-matched controls (non-carriers). More specifically, possible differences in the breast tissue at time of enrollment into the study (reflecting changes potentially occurring in adolescence) and in the rate of breast tissue change over time (reflecting rate of tissue transformation from normal to ultimately malignant state). The overall goal is to develop a pre-screening technique to survey or monitor the risk of breast tissue and to advise the earliest point when imaging techniques (e.g. MRI) should be initiated or when more drastic primary prevention measures are recommended.

ELIGIBILITY:
Inclusion Criteria:

BrCa carriers (cases)

* Attending one of the three participating high-risk screening centres
* Confirmed BrCa1 or BrCa2 mutation status through genetic testing

High-Risk (cases)

* Attending one of the three participating high-risk screening centres
* Confirmed negative BrCa1/2 status through genetic testing

BrCa non-carriers (controls)

* Attain a GAIL model score of <1.1 and have <10% risk of carrying the BRCa mutation Determined by the Penn II model)
* Controls from high-risk screening centre with confirmed BrCa1/2 negative status through genetic testing
* Preference will be given to sisters or first degree cousins of BrCa carriers

Exclusion Criteria:

Cases and Controls

* Prior diagnosis or Breast or Ovarian Cancer
* Bilateral biopsy or fine needle aspiration within 1 year of study start
* Bilateral mastectomy, lumpectomy or cosmetic alteration (reduction/augmentation)
* Previous or current chemotherapy or prevention therapy (Tamoxifen)
* Less than 3 years post pregnancy at study start
* inability to provide informed consent due to language or cognitive difficulties

  *For controls only
* Family history of breast cancer where family member had an early diagnosis (before age 45 years)
* Family history or ovarian cancer

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases are recruited from three participating high-risk screening centres: Familial Breast and Ovarian Cancer Programs at Mount Sinai Hospital and/or Princess Margaret Hospital (Toronto, Ontario, Canada), the Juravinski Cancer Center (Hamilton, Ontario, Canada) and Women's College Hsopital (toronto, Ontario, Canada). Controls are recruited from the respective geographical locations.
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2009-10; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Difference in rate of change between the high risk groups and the respective controls | over the 4 year duration of the study
  the primary optical measurements are utilized to determine principal component scores in the analysis which in turn will be used as time dependent variable in a linear regression analysis to determine the rate of change.

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Lilge, PhD, Principal Investigator — Ontario Cancer Institute, University Health Network, Toronto, Ontario, Canada M5G 2M9; Department of Biophysics and Bioimaging, University of Toronto, Toronto, Ontario, Canada M5G 2M9
Locations (4):
- Canada (4):
  - Juravinski Cancer Center, Hamilton Health Sciences, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Blyschak K, Simick M, Jong R, Lilge L. Classification of breast tissue density by optical transillumination spectroscopy: optical and physiological effects governing predictive value. Med Phys. 2004 Jun;31(6):1398-414. doi: 10.1118/1.1738191. PMID 15259643
- [Background] Simick MK, Jong R, Wilson B, Lilge L. Non-ionizing near-infrared radiation transillumination spectroscopy for breast tissue density and assessment of breast cancer risk. J Biomed Opt. 2004 Jul-Aug;9(4):794-803. doi: 10.1117/1.1758269. PMID 15250768
- [Background] Blackmore KM, Knight JA, Jong R, Lilge L. Assessing breast tissue density by transillumination breast spectroscopy (TIBS): an intermediate indicator of cancer risk. Br J Radiol. 2007 Jul;80(955):545-56. doi: 10.1259/bjr/26858614. Epub 2007 May 30. PMID 17537757
- [Background] Simick MK, Lilge L. Optical transillumination spectroscopy to quantify parenchymal tissue density: an indicator for breast cancer risk. Br J Radiol. 2005 Nov;78(935):1009-17. doi: 10.1259/bjr/14696165. PMID 16249602